CLINICAL TRIAL: NCT05456867
Title: A Multi-center, Non-interventional, Prospective Study of Durvalumab in Unresectable Locally Advanced NSCLC in Routine Clinical Practice in Russia
Acronym: NIS durvalumab
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4194R00027
Record Dates: First submitted 2022-05-26; First posted 2022-07-13 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: NSCLC, Non-small-cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
Durvalumab was approved in the Russian Federation for use after both concurrent and subsequent CRT until disease progression. Currently, there is no real-world data regarding the safety and real world effectiveness of durvalumab in this indication. Moreover, generation data on the safety and real world effectiveness of durvalumab after concurrent chemo-radiation therapy (cCRT) and subsequent chemo-radiation therapy (sCRT) in routine practice in the Russian Federation will be of high relevance.

The other important question that needs to be addressed is the duration of treatment with durvalumab and its' influence on the relevant outcomes. According to the Russian label, it is possible to continue treatment with durvalumab until disease progression, although current data from the PACIFIC trial provide the results on 12 months duration of durvalumab treatment. The real-world data about the duration of treatment with durvalumab in the Russian population and its' influence on various outcomes would be very important.

Among other goals, the current study is aimed to analyze factors influencing the effectiveness of durvalumab therapy in the real-world setting (e.g. duration of treatment, delays in the start of treatment with durvalumab after CRT over, early discontinuation due to any factors including AEs, etc.). The study also aims to elucidate treatment approaches after discontinuation from durvalumab (post-progression outcomes and treatment in case of discontinuation due to AEs). This study will support the understanding of described factors and will take and an attempt to optimize the treatment process to improve outcomes for patients

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if all of the following inclusion criteria and none of the exclusion criteria apply:

* Written informed consent obtained from the patient prior to performing any protocol-related procedures
* Age ≥18 years at time of study entry
* Patients must have histologically or cytologically documented diagnosis of NSCLC with a locally advanced, or locally recurrent, unresectable (stage III) disease (according to American Joint Committee on Cancer [AJCC] lung cancer edition 8)
* Patients must have completed a platinum-based chemotherapy with radiation therapy (concurrent or sequential) without evidence of disease progression
* Patients must have been treated with at least one dose of durvalumab

Exclusion Criteria:

Any subject who meets any of the following criteria will not qualify for entry into the study:

* Absence or missing of written informed consent form
* Patients treated with durvalumab in clinical studies
* Absence of essential data to obtain all necessary information
* Confirmation that the subject was already included in this study before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study may include all patients who have received the first dose of durvalumab prior to study participation.
  To enter in the study, patients must have completed a platinum-based chemotherapy concurrently or sequentially with radiation therapy without evidence of disease progression. There is no fixed maximum duration for durvalumab treatment. Treatment with durvalumab continues until the physician determines that it is in the patient's best interest to stop therapy.
  It is expected to recruit 300 patients from approximately 25 cites.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety of durvalumab in patients with unresectable locally advanced NSCLC without progression after CRT in routine practice of the Russian Federation. | Up to 54 month
Number of any treatment (durvalumab) related AEs by physician diagnosis within all treatment period plus 3 months after durvalumab discontinuation. | Up to 54 month
Number of any treatment (durvalumab) related AEs by physician diagnosis within all treatment period plus 3 months after durvalumab discontinuation separately for fix dose (1500mg every 4 weeks) and 10mg/kg every 2 weeks dosage. | Up to 54 month
Number of irAEs | Up to 54 month
Number of SAEs | Up to 54 month
Number of grade 3-4 AEs | Up to 54 month
Number of post discontinuation irAEs | Up to 54 month
Number of AESIs | Up to 54 month
Number of AEs which lead to discontinuation | Up to 54 month
Time to pneumonitis [median, months] | Up to 54 month
Distribution of pneumonitis grades | Up to 54 month
Nature of pneumonitis by physician diagnosis [radiation or immune-related] | Up to 54 month
Duration of pneumonitis [median, months] | Up to 54 month

CONTACTS AND LOCATIONS:
Locations (24):
- Russia (24):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Grozny
  - Research Site, Irkutsk
  - Research Site, Kemerovo
  - Research Site, Khanty-Mansiysk
  - Research Site, Kostroma
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, N.Novgorod
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Sochi
  - Research Site, Surgut
  - Research Site, Syktyvkar
  - Research Site, Tomsk
  - Research Site, Ufa
  - Research Site, Vologda
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
  - Research Site, Yuzhno-Sakhalinsk